CLINICAL TRIAL: NCT00901290
Title: A Randomized, Open-Label, Two-way Crossover Study to Determine the Effects of Co-administration of AZD7325 and a Monophasic Oral Contraceptive Containing Ethinyl Estradiol and Norgestimate in Healthy Female Subjects
Brief Title: Determine the Effects of C-administration of AZD7325 and an Oral Contraceptive in Healthy Female Subjects
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: suspended pending data analysis
Sponsor: AstraZeneca (Industry)
Responsible Party: MSD, AstraZeneca
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: D1140C00018
Record Dates: First submitted 2009-05-12; First posted 2009-05-13 (Estimated); Last update posted 2010-12-10 (Estimated); Status verified 2009-10

CONDITIONS: Pharmacokinetics
Keywords: oral contraceptive
MeSH Terms: interventions — Moxifloxacin; 4-amino-8-(2-fluoro-6-methoxy-phenyl)-N-propylcinnoline-3-carboxamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): monophasic oral contraceptive
  Interventions: Drug: monophasic oral contraceptive
- 2 (Experimental): AZD7325
  Interventions: Drug: AZD7325

INTERVENTIONS:
Drug: monophasic oral contraceptive — mg, oral dose
  Other Names: ORTHO-CYCLEN
  Arms: 1
Drug: AZD7325 — mg, oral dose
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate the effect of repeated doses of AZD7325 on the pharmacokinetics of ORTHO-CYCLEN, a monophasic oral contraceptive

ELIGIBILITY:
Inclusion Criteria:

* If previously pregnant, must be > 6 month post-partum at the time of randomization
* Body Mass Index (BMI) greater than or equal to 18 and less than or equal to 30 kg/m2

Exclusion Criteria:

* Use of any prescription medication within 14 days of screening
* current smoker or history of smoking within the last 3 months prior to enrollment
* Abnormal pap smear exam result within one year of enrollment.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Estimated)
Dates: Start 2009-05; Primary Completion 2009-09 (Estimated); Study Completion 2009-09 (Estimated)

PRIMARY OUTCOMES:
To evaluate the effect of repeated doses of AZD7325 on the pharmacokinetics of ORTHO-CYCLEN | weekly

SECONDARY OUTCOMES:
Characterize the pharmacokinetics of progesterone, luteinizing hormone, follicle-stimulating hormone, and sex hormone binding globulin following dosing with monophasic oral contraceptive (ORTH-CYCLEN) alone and following co-administration with AZD7325 | weekly
To characterize the steady-state pharmacokinetics of AZD7325 | weekly
To examine the safety and tolerability of AZD7325 in combination with the monophasic oral contraceptive (ORTHO-CYCLEN) | weekly

CONTACTS AND LOCATIONS:
Overall Officials: Eleanor Lisbon, MD, MPH, Principal Investigator — Quintiles Phase I Services
Locations (1):
- Research Site, Overland Park, Kansas, United States